CLINICAL TRIAL: NCT05025995
Title: Can Garfield Make Children Eat Healthier? A Cluster-randomized Controlled Trial to Examine the Effect of a Serious Health Game on Children's Eating Behavior
Brief Title: The Effect of a Serious Health Game on Children's Eating Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Responsible Party: Principal Investigator, Frans Folkvord, Assistant professor, Tilburg University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BSI-01
Record Dates: First submitted 2021-08-03; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious health game (Experimental): Children played a serious health game with Garfield promoting health behavior, such as less intake of energy dense snacks, drink more water, and exercise more often.
  Interventions: Behavioral: Serious health game
- control (Experimental): Children in this condition did not play a serious health game and were in control condition.
  Interventions: Behavioral: Serious health game

INTERVENTIONS:
Behavioral: Serious health game — Serious health game

SUMMARY:
Background: Currently the dietary intake patterns of children do not meet the prescribed dietary guidelines. Consequently childhood obesity is one of the most serious health concerns. Therefore, innovative methods need to be developed and tested in order to effectively improve the dietary intake of children. Learning children how to cope with the overwhelming number of unhealthy food cues could be conducted effectively by serious health games.

Objective: The main aim of this study was to examine the effect of a serious health computer game on young children's eating behavior and attitudes towards healthy and unhealthy foods.

Methods: A cluster-randomized controlled trial with a between-subject design was conducted (N=157; 8-12 years), whereby children played a game that promoted a healthy lifestyle or were in the control condition. Children in the control condition attended regular classes and did not play a game. The game was designed in collaboration with researchers and pilot-tested before conducting the experiment among a group of children repeatedly. After one week of playing, attitudes towards food snacks and actual intake was assessed, whereby children could eat at libitum from fruits or energy-dense snacks.

ELIGIBILITY:
Inclusion Criteria:

* primary school between group 5 and 8

Exclusion Criteria:

* n.a.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
calorie intake of energy dense snacks (candy) and fruits (bananas and apples) | 1 week after treatment
  Energy dense snacks and fruits

CONTACTS AND LOCATIONS:
Locations (1):
- Tilburg School of Humanities and Digital Sciences, Tilburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Folkvord F, Haga G, Theben A. The Effect of a Serious Health Game on Children's Eating Behavior: Cluster-Randomized Controlled Trial. JMIR Serious Games. 2021 Sep 2;9(3):e23050. doi: 10.2196/23050. PMID 34473061